CLINICAL TRIAL: NCT03490513
Title: Aromatase Inhibitors and Weight Loss in Severely Obese Men With Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Reina Villareal MD, Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-41814
Record Dates: First submitted 2018-03-22; First posted 2018-04-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Hypogonadism, Hypogonadotropic; Obesity
MeSH Terms: conditions — Hypogonadism; Obesity | interventions — Anastrozole

STUDY DESIGN:
Intervention Model Description: Intervention: Subjects will be randomized to 2 groups: 1) placebo+weight loss, and 2) anastrozole+weight loss. Intervention will be conducted for 12 months.
  Weight loss + placebo: Subjects will participate in a supervised dietary and exercise program plus a placebo.
  Anastrozole + weight loss: Subjects will participate in a supervised dietary and exercise program plus the aromatase inhibitor, anastrozole at 1 mg daily.
  All subjects will be provided supplements to ensure an intake of ~1500 mg of calcium/day and ~1000 IU vitamin D/day. We will maintain a serum 25-hydroxyvitamin D level of at least 30 ng/dl. Additional vitamin D supplements will be provided for those with level <30 ng/dl.
  Dosage adjustments and monitoring will be done by an unblinded investigator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One of the investigators will be unblinded for safety purposes and to adjust the dose of medication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Weight loss plus placebo (Placebo Comparator): Participants will take a placebo every day, attend behavioral classes conducted by a dietitian, receive instruction on how to loss 10% of their body weight and undergo supervised exercise training program.
  Interventions: Drug: Placebo
- Weight loss plus anastrozole (Experimental): Participants will take Anastrozole 1mg per day, attend behavioral classes conducted by a dietitian, receive instruction on how to loss 10% of their body weight and undergo supervised exercise training program.
  Interventions: Drug: anastrozole (1 mg/day)

INTERVENTIONS:
Drug: anastrozole (1 mg/day) — Participants will take Anastrozole 1mg per day, attend behavioral classes conducted by a dietitian, receive instruction on how to loss 10% of their body weight and participate in a supervised exercise training program.
  Other Names: Weight loss
  Arms: Weight loss plus anastrozole
Drug: Placebo — Participants will take a placebo tablet every day, attend behavioral classes conducted by a dietitian, receive instruction on how to loss 10% of their body weight and participate in a supervised exercise training program.
  Other Names: Weight loss
  Arms: Weight loss plus placebo

SUMMARY:
The investigators have preliminary data suggesting that obese patients with hypogonadotropic hypogonadism (HHG) have minimal benefit from testosterone therapy likely because of its conversion to estradiol by the abundant aromatase enzyme in the adipocytes. The increased conversion of androgens into estrogens in obese men results in a negative feedback of high estradiol levels on hypothalamus and pituitary, inhibiting the production of gonadotropin-releasing hormone (GnRH), luteinizing hormone (LH) and follicle stimulating hormone (FSH) and, as a consequence, of testosterone by the testis. Testosterone administration could increase estradiol production, further promoting the inhibitory feedback to the hypothalamic-pituitary-gonadal axis. Although weight loss from lifestyle modification has been shown to reduce estradiol and increase testosterone levels, the effect is at best modest and weight regain results in recurrence of hypogonadism. The use of aromatase inhibitors, in combination with weight loss, could be an effective alternative strategy due to its action at the pathophysiology of the disease.

Intervention Subjects (body mass index of ≥35, testosterone <300 ng/dl) will be randomized to the active (anastrozole) or control (placebo) group. Anastrozole 1 mg tablet / day will be self-administered with or without food, at around the same time every day (active group); placebo 1 tablet/day with or without food to take at around the same time every day (control group). The study duration will be 12 months.

Both groups will undergo lifestyle intervention consisting of diet and supervised exercise program. Target weight loss will be at least 10% of baseline body weight during the intervention. Subjects will attend weekly group behavior modification sessions which will last ~75-90 min for the first 3 months and decreased to every two weeks from 3 to 12 months. Subjects will attend supervised research center-based exercise sessions during the first 6 months followed by community fitness center-based sessions during the next 6 months for at least 2 d/wk, with recording of home-based exercises for the other 2-4 days/week.

Although the above original protocol requires the participants to come to our center for dietary and exercise training, since the Covid19 pandemic, study participants were given the following options for lifestyle intervention: 1) in-person visits at our facility for dietary classes and exercise training, 2) to enlist in the gym of their choice with membership paid for by the study, or 3) virtual method of lifestyle intervention. These amendments were put in place due to Covid 19 restrictions; however, we decided to keep these methods because most of our subjects prefer them over coming for in-person visits at our lab even after COVID restrictions were lifted. Since the study had just the first 25 subjects enrolled prior to COVID outbreak, majority of the subject's lifestyle interventions were done by virtual dietary classes every week for the first 3 months and then every 2 weeks thereafter either as a group or by one-on-one sessions. Exercise program was also supervised by exercise physiologist virtually or by phone for subjects who want to exercise at a community gym

DETAILED DESCRIPTION:
After age of 40, testosterone (T) production in men gradually decreases at a rate of 1.6% per year for total and to 2-3% per year for bioavailable T. This reduction in T production in men parallels the age-associated loss of muscle mass that leads to sarcopenia and impairment of function and the age-associated loss of bone mass that leads to osteopenia and fracture risk.

Hypogonadism is a condition associated with multiple symptom complex including fatigue, depressed mood, osteoporosis, gain of fat mass, loss of libido and reduced muscle strength, all of which deeply affect patient quality of life. The prevalence of hypogonadism among obese men was estimated to be as much as 40% and could as much as 50% if they are also diabetic, with levels of androgens decreasing proportionately to the degree of obesity.

In obese men, the age-related decline in T is exacerbated by the suppression of the hypothalamic-pituitary-gonadal axis by hyperestrogenemia. The high expression of aromatase enzyme in the adipose tissue enhances the conversion of androgens into estrogens which in turn exerts a negative feedback on hypothalamus and pituitary, inhibiting the production of gonadotropin-releasing hormone (GnRH), luteinizing hormone (LH) and follicle stimulating hormone (FSH) and, as a consequence, of T by the testis resulting in hypogonadotropic hypogonadism (HH). Considering the high aromatase expression in the adipose tissue, the administration of T among obese men with HHG could increase the conversion of the substrate T to estradiol (E2) and fuels the negative feedback on hypothalamus and pituitary, producing a greater suppression of GnRH and gonadotropins. Thus, men with obesity induced HHG may benefit from other treatment strategies that target the pathophysiology of the disease.

Although weight loss intervention improves hormonal and metabolic abnormalities related to obesity, the increase in T levels induced by weight loss are often lost due to weight regain, which is very frequent among patients undergoing massive weight loss. One possible approach is the use of aromatase inhibitors (AI) to stop the conversion of T to E2 thereby interrupting the vicious cycle of E2 inhibition of the hypothalamic-pituitary-gonadal axis and restoring T production to normal levels. Since weight loss remains the standard of care for obese patients, the investigators propose the following OBJECTIVES:

1. To evaluate the effect of an AI plus WL (AI+WL) compared to WL alone on the changes in hormonal profile in severely obese men with HHG.
2. To evaluate the effect of an AI+WL compared to WL alone on the changes in muscle strength and muscle mass, and symptoms of hypogonadism in severely obese men with HHG.
3. To evaluate the effect of an AI+WL compared to WL alone on the changes in body composition and metabolic risk factors in severely obese men with HHG.
4. To evaluate the effect of an AI+WL compared to WL alone on the changes in bone mineral density (BMD), bone markers, and bone quality in severely obese men with HHG.

As secondary aim, the investigators will elucidate the mechanism for the anticipated positive effects of AI+WL on obesity-associated HHG.

This is a randomized double-blind placebo-controlled study comparing the effect of weight loss + anastrozole to weight loss + placebo for 12 months on the hormonal profile and symptoms associated with hypogonadism in severely obese men with a body mass index (BMI) of more or equal to 35 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* obese men with body mass index (BMI) of ≥35 kg/m2
* age between 40 to 65 years old
* average fasting testosterone level from 2 measurements taken between 8 to 10 AM on 2 separate days of <300 ng/dl
* Luteinizing Hormone (LH) of <9.0 mIU/L
* Estradiol of ≥17 pg/ml
* Symptoms consistent with androgen deficiency as assessed by Androgen Deficiency in Aging Male (ADAM) questionnaire

Exclusion criteria:

* pituitary or hypothalamic disease,
* drugs affecting gonadal hormone levels, production and action or bone metabolism (bisphosphonates, teriparatide, denosumab, glucocorticoids, phenytoin)
* diseases affecting bone metabolism (e.g. hyperparathyroidism, untreated hyperthyroidism, osteomalacia, chronic liver disease, significant renal failure, hypercortisolism, malabsorption, immobilization, Paget's disease),
* prostate carcinoma or elevated serum prostate specific antigen (PSA)> 4 ng/ml,
* Hematocrit > 50%,
* untreated severe obstructive sleep apnea,
* Cardiopulmonary disease (e.g. recent myocardial infarction, unstable angina, stroke) or unstable disease (e.g., New York Heart Association Class III or IV congestive heart failure
* severe pulmonary disease requiring steroid pills or the use of supplemental oxygen (that would contraindicate exercise or dietary restriction)
* History of deep vein thrombosis or pulmonary embolism
* severe lower urinary tract or prostate symptoms with International Prostate Symptom Score (IPSS) above 19
* excessive alcohol or substance abuse
* unstable weight (i.e. >±2 kg) in the last 3 months
* condition that could prevent from completing the study
* screening bone mineral density (BMD) T-score of <-2.0 at the spine, femoral neck or total femur
* history of osteoporosis or fragility fracture
* Diabetes mellitus with a fasting blood glucose of >140 mg/dl, and/or Hemoglobin A1C (A1C) >8.5%.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is investigating obesity induced male hypogonadism
Enrollment: 121 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Hormonal Profile Changes | 12 months
  Assessed by changes in serum testosterone levels.
Changes in muscle strength | 12 months
  Assessed by changes in knee extension strength using a dynamometer.
Changes in Lean mass | 12 months
  Assessed by body composition tissue measurement using dual energy x-ray absorptiometry.
Changes in total hip bone mineral density (BMD) | 12 months
  Assessed by dual energy absorptiometry.

SECONDARY OUTCOMES:
Other gonadal hormone | 12 months
  Assessed by changes in serum estradiol
Pituitary hormone | 12 months
  Assessed by changes in serum luteinizing hormone (LH)
Pituitary hormone | 12 months
  Assessed by changes in serum follicle stimulating hormone (FSH)
Changes in thigh muscle volume | 12 months
  Assessed magnetic resonance imaging of both thighs.
Changes in symptoms of hypogonadism | 12 months
  Assessed by the Androgen Deficiency in Aging Male (ADAM) questionnaire; higher scores indicating worse outcome
Changes in symptoms of hypogonadism | 12 months
  Assessed by the International Index of Erectile Function (IIEF) questionnaire; higher scores indicating better outcome
Changes in symptoms of hypogonadism | 12 months
  Assessed by the 36-Item Short-Form Health Survey (SF-36) questionnaire; scores on the physical and mental component subscales of the SF-36 range from 0 to 100, with higher scores indicating better health status
Changes in visceral adipose tissues | 12 months
  Assessed by dual energy x-ray absorptiometry
Changes in metabolic risk factors | 12 months
  Assessed by hemoglobin A1C
Changes in metabolic risk factors | 12 months
  Assessed by lipid profile
Changes in metabolic risk factors | 12 months
  Assessed by homeostasis model assessment for insulin resistance (HOMA-IR)
Changes in volumetric bone density | 12 months
  Assessed by high-resolution peripheral quantitative computer tomography
Changes in bone quality | 12 months
  Assessed by changes in finite element analysis using high-resolution peripheral quantitative computer tomography
Changes in bone markers | 12 months
  Assessed by serum C-telopeptide
Changes in bone markers | 12 months
  Assessed by serum osteocalcin
Changes in bone markers | 12 months
  Assessed by serum procollagen 1 Intact N-terminal

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VAMC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schneider G, Kirschner MA, Berkowitz R, Ertel NH. Increased estrogen production in obese men. J Clin Endocrinol Metab. 1979 Apr;48(4):633-8. doi: 10.1210/jcem-48-4-633. PMID 429508
- [Result] Corona G, Rastrelli G, Monami M, Saad F, Luconi M, Lucchese M, Facchiano E, Sforza A, Forti G, Mannucci E, Maggi M. Body weight loss reverts obesity-associated hypogonadotropic hypogonadism: a systematic review and meta-analysis. Eur J Endocrinol. 2013 May 2;168(6):829-43. doi: 10.1530/EJE-12-0955. Print 2013 Jun. PMID 23482592
- [Result] Armamento-Villareal R, Aguirre LE, Qualls C, Villareal DT. Effect of Lifestyle Intervention on the Hormonal Profile of Frail, Obese Older Men. J Nutr Health Aging. 2016 Mar;20(3):334-40. doi: 10.1007/s12603-016-0698-x. PMID 26892583
- [Result] Feldman HA, Longcope C, Derby CA, Johannes CB, Araujo AB, Coviello AD, Bremner WJ, McKinlay JB. Age trends in the level of serum testosterone and other hormones in middle-aged men: longitudinal results from the Massachusetts male aging study. J Clin Endocrinol Metab. 2002 Feb;87(2):589-98. doi: 10.1210/jcem.87.2.8201. PMID 11836290
- [Result] Khosla S, Melton LJ 3rd, Atkinson EJ, O'Fallon WM. Relationship of serum sex steroid levels to longitudinal changes in bone density in young versus elderly men. J Clin Endocrinol Metab. 2001 Aug;86(8):3555-61. doi: 10.1210/jcem.86.8.7736. PMID 11502778
- [Result] Bassil N, Alkaade S, Morley JE. The benefits and risks of testosterone replacement therapy: a review. Ther Clin Risk Manag. 2009 Jun;5(3):427-48. doi: 10.2147/tcrm.s3025. Epub 2009 Jun 22. PMID 19707253
- [Result] Kaplan SA, Lee JY, O'Neill EA, Meehan AG, Kusek JW. Prevalence of low testosterone and its relationship to body mass index in older men with lower urinary tract symptoms associated with benign prostatic hyperplasia. Aging Male. 2013 Dec;16(4):169-72. doi: 10.3109/13685538.2013.844786. Epub 2013 Oct 17. PMID 24134648
- [Result] Dhindsa S, Miller MG, McWhirter CL, Mager DE, Ghanim H, Chaudhuri A, Dandona P. Testosterone concentrations in diabetic and nondiabetic obese men. Diabetes Care. 2010 Jun;33(6):1186-92. doi: 10.2337/dc09-1649. Epub 2010 Mar 3. PMID 20200299
- [Result] Giagulli VA, Kaufman JM, Vermeulen A. Pathogenesis of the decreased androgen levels in obese men. J Clin Endocrinol Metab. 1994 Oct;79(4):997-1000. doi: 10.1210/jcem.79.4.7962311.
- [Result] Strain GW, Zumoff B, Kream J, Strain JJ, Deucher R, Rosenfeld RS, Levin J, Fukushima DK. Mild Hypogonadotropic hypogonadism in obese men. Metabolism. 1982 Sep;31(9):871-5. doi: 10.1016/0026-0495(82)90175-5. PMID 6811834
- [Derived] Joad S, Ballato E, Deepika F, Gregori G, Fleires-Gutierrez AL, Colleluori G, Aguirre L, Chen R, Russo V, Fuenmayor Lopez VC, Qualls C, Villareal DT, Armamento-Villareal R. Hemoglobin A1c Threshold for Reduction in Bone Turnover in Men With Type 2 Diabetes Mellitus. Front Endocrinol (Lausanne). 2021 Dec 28;12:788107. doi: 10.3389/fendo.2021.788107. eCollection 2021. PMID 35027909
- [Derived] Vigevano F, Gregori G, Colleluori G, Chen R, Autemrongsawat V, Napoli N, Qualls C, Villareal DT, Armamento-Villareal R. In Men With Obesity, T2DM Is Associated With Poor Trabecular Microarchitecture and Bone Strength and Low Bone Turnover. J Clin Endocrinol Metab. 2021 Apr 23;106(5):1362-1376. doi: 10.1210/clinem/dgab061. PMID 33537757